CLINICAL TRIAL: NCT00862485
Title: MCA Doppler Studies in Neborns Following Exchange Transfusion
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, wamir, MD, Rambam Health Care Campus
Other Study IDs: 1910CTIL
Record Dates: First submitted 2009-03-15; First posted 2009-03-17 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Exchange Transfusion

STUDY DESIGN:
Observational Model: Case-Only

GROUPS / COHORTS (1):
- StudyGroup

SUMMARY:
The purpose of this study is to study MCA Doppler before and after exchange transfusion in newborns.

ELIGIBILITY:
Inclusion Criteria:

* Newborns who need exchange transfusion by accepted criteria

Max Age: 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: newborns
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-03; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Doppler measurement | one year
  Doppler of middle cerebral artery

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel